CLINICAL TRIAL: NCT05118087
Title: Comparison of Bracing With Co-aptation Splinting for the Initial Treatment of Acute Humeral Shaft Fractures: The COBRAS Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-00438
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Humeral Fractures
Keywords: Sarmiento Brace; Coaptation Splint
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coaptation Splint (Active Comparator)
  Interventions: Procedure: Webril Padded Plaster Splint
- Sarmiento Brace (Active Comparator)
  Interventions: Procedure: Pre-Fabricated Fracture Brace

INTERVENTIONS:
Procedure: Webril Padded Plaster Splint — Patients in the coaptation splint group will have a webril padded plaster splint that is placed around the humerus. The forearm and wrist are then suspended in a cuff and collar.
  Arms: Coaptation Splint
Procedure: Pre-Fabricated Fracture Brace — Patients in the sarmiento group will be given a fitted pre-fabricated fracture brace with a cuff and collar for the forearm. The patients will be educated on brace maintained, tightening, and care during at the time of the ER encounter.
  Arms: Sarmiento Brace

SUMMARY:
The goal of this study is to determine which initial method of immobilization for humeral shaft fractures in the emergency room maximizes patient comfort. The two methods of initial management for humeral shaft fractures are sarmiento bracing (pre-fabricated fracture brace) and coaptation splinting. In this study, the team will compare patient related outcomes and comfort for each method of initial management of humeral shaft fractures. Participant pain, narcotic usage, and function will be tracked over a 2 week period to see which method of immobilization is preferred.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting to an emergency room or ICARE in the participating centers with an acute humeral shaft fracture
2. Age above 18 and skeletally mature
3. Isolated Injury
4. Treated non-operatively first 2 weeks

Exclusion Criteria:

1. Open fractures
2. Poly trauma
3. Injuries deemed operative by attending surgeon
4. Patients undergoing treatment for malignancy
5. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Score on Pain Visual Analogue Scale (VAS) | Week 1 post-treatment
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. The total range of score is 0 (no pain) to 10 (unbearable pain); the higher the pain, the greater the amount of pain.
Score on Pain Visual Analogue Scale (VAS) | Week 2 post-treatment
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. The total range of score is 0 (no pain) to 10 (unbearable pain); the higher the pain, the greater the amount of pain.
Number of Tramadol Pills Taken | Week 1 post-treatment
  All patients will be discharged with 28 pills of tramadol 50mg. At week 1 follow-up, number of tramadol pills taken will be reported.
Number of Tramadol Pills Taken | Week 2 post-treatment
  All patients will be discharged with 28 pills of tramadol 50mg. At week 2 follow-up, number of tramadol pills taken will be reported.

SECONDARY OUTCOMES:
Incidence of cutaneous complications | Week 2 post-treatment
  Cutaneous complications between immediate fracture bracing and coaptation splints in the ER within the first 2 weeks of treatment will be reported
Score on PROMIS - Physical Function - Short Form 10b | Week 1 post-treatment
  PROMIS consists of 10 statements/questions that are scored 1-5 each. The total range of score is 10-50; a higher score indicates less difficulty performing an activity.
Score on PROMIS - Physical Function - Short Form 10b | Week 2 post-treatment
  PROMIS consists of 10 statements/questions that are scored 1-5 each. The total range of score is 10-50; a higher score indicates less difficulty performing an activity.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Ganta, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Winthrop Hospital, Garden City, New York
  - NYU Langone Health, New York, New York
  - Jamaica Hospital Medical Center, Queens, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to abhishek.ganta@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.